CLINICAL TRIAL: NCT02471261
Title: Elastography as Gouty Arthropathy Outcome (EGO), a Pilot Study.
Brief Title: Elastography as Gouty Arthropathy Outcome (EGO)
Status: Completed | Type: Observational
Sponsor: Arthritis & Rheumatism Associates, P.C. (Other)
Responsible Party: Sponsor
Other Study IDs: ESR-14-10146
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Elastography as Gouty Arthropathy Outcome (EGO), a pilot study.

DETAILED DESCRIPTION:
Pilot study to assess 10 subjects with tophaceous gout on urate lowering therapy or about to begin urate lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are at least 18 years of age but younger than or equal to 99 years of age.
2. Subjects with gouty arthritis as determined by the ACR 1977 classification criteria for gouty arthritis.
3. Subjects with one palpable tophus detectable by one of the three clinical parameters described.

   -

Exclusion Criteria:

1. Subjects who are not eligible for urate lowering treatment or show a hypersensitivity to these drugs or class of compounds.
2. Subjects with significant cardiovascular, neuropsychiatric, hematologic, hepatic, renal or endocrine dysfunction who in the opinion of the principal investigator are unfit for participation in a clinical trial.
3. Subjects for which the clinical and laboratory assessment would provide undue discomfort and / or are contraindicated.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A pilot study to assess 10 subjects with tophaceous gout on urate lowering therapy or about to begin urate lowering therapy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Elastography as Gouty Arthropathy Outcome (EGO), a pilot study | 1 year
  Observational trial to measure gouty arthritis changes in subject taking urate lowering therapies

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Rheumatology and Bone Research, Wheaton, Maryland, United States